CLINICAL TRIAL: NCT02363153
Title: A Pilot Study of Diet and Exercise Therapy in Pompe Disease
Brief Title: Diet and Exercise in Pompe Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201400844
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Pompe Disease; Glycogen Storage Disease Type II; Lysosomal Storage Diseases
MeSH Terms: conditions — Glycogen Storage Disease Type II; Lysosomal Storage Diseases | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diet and Exercise (Experimental): Patients will be given an individualized diet and exercise plan by a physical therapist and registered dietician. The diet and exercise plan will be carried out by the participant for 16 weeks. The exercise plan, an aerobic and strength training regimen, will be performed under the supervision of a personal trainer or certified exercise physiologist that is local to the participant. The participant will complete core-stabilizing exercises which can be performed at home or in an approved group class. The participant will wear an activity tracker at all times during this 16 week period, and will be asked to manually enter data into a phone app, such as daily food intake and weight.
  Interventions: Other: Diet and Exercise

INTERVENTIONS:
Other: Diet and Exercise — Exercise will consist of 2x/week aerobic exercise, 2x/week strength training and 1x/week core-stabilizing exercise.
  Diet will be constructed so that 30% of the daily caloric goal will be protein, 35% fat, and 35% carbohydrates.

SUMMARY:
This study examines the effects of individualized diet and exercise plans on muscle strength, quality of life and respiratory function in Pompe disease. Subjects will be given a diet and exercise plan based on their individual needs, which will be followed for 16 weeks. Participants will also be provided with an activity tracker in order to track their exercise activities, access to an app that will allow them to input their daily food intake, and they will also come to the University of Florida for exercise tests, respiratory tests and questionnaires.

DETAILED DESCRIPTION:
Pompe is a rare disease, which occurs in approximately 1 in 40,000 births. It is a progressive and often fatal neuromuscular disorder resulting from a mutation in the gene for acid alpha- glucosidase (GAA), an enzyme necessary for the degradation of glycogen. Common symptoms include skeletal and smooth muscle myopathy, resulting in respiratory insufficiency, peripheral muscle weakness and generalized fatigue.

The progressive myopathy in Pompe disease seems to be influenced by increased muscle protein breakdown. The increased muscle protein breakdown leads to muscle wasting, weakness, increased resting energy expenditure and, consequently, increased fatigue. Our hypothesis is that a high protein, low carbohydrate diet associated with regular physical exercise will improve respiratory and peripheral muscle functions in Pompe disease.

In this study, we will investigate the effects of 16 weeks of planned diet and exercise in adolescent and young adult (15-55 years old) individuals with Pompe disease using an activity tracker.

The participant will be asked to come to the University of Florida 4 times throughout the study (screening, baseline, +/- 15 days of completing the diet and exercise plan and a follow up three months later) for exercise testing, quality of life questionnaires, respiratory function testing and blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 15-55 years of age;
* Have a diagnosis of Pompe disease, as defined by protein assay and/or DNA sequence of the acid alpha-glucosidase gene, with present clinical symptoms of the disease;
* Be naïve to ERT or receiving ERT for at least eighteen months prior to beginning study;
* Be able to walk at least 40m in the 6 minute walk test.
* Willing to comply with study requirements

Exclusion Criteria:

* Be pregnant;
* Be in the lower limit for pulmonary function; FVC < 30% predicted;
* Be dependent on assisted ventilation;
* Be dependent on wheelchair;
* Have evidence of clinical heart failure;
* Have any contraindication to exercise

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Change in results of Brief Patient-Reported Outcomes Quality of Life (PROQOL) | Baseline, Month 4
  The PROQOL assesses quality of life and health status to improve patient care
Change in FVC | Baseline, Month 4
  Forced Vital Capacity (FVC) is the amount of air that can be forcefully exhaled after a full inspiration, and is an indicator of overall respiratory function
Change in overall QMT score | Baseline, Month 4
  Quantitative muscle testing (QMT) measures peripheral muscle strength

SECONDARY OUTCOMES:
Compliance to diet and exercise plans | Month 4
  Patients will be evaluated on their compliance to the diet and exercise plan they are assigned, by comparing activities assigned vs. activities completed

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Corti, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Clinical Research Center, Gainesville, Florida, United States

REFERENCES:
- [Background] Bodamer OA, Leonard JV, Halliday D. Dietary treatment in late-onset acid maltase deficiency. Eur J Pediatr. 1997 Aug;156 Suppl 1:S39-42. doi: 10.1007/pl00014270. PMID 9266214
- [Background] van der Ploeg AT, Clemens PR, Corzo D, Escolar DM, Florence J, Groeneveld GJ, Herson S, Kishnani PS, Laforet P, Lake SL, Lange DJ, Leshner RT, Mayhew JE, Morgan C, Nozaki K, Park DJ, Pestronk A, Rosenbloom B, Skrinar A, van Capelle CI, van der Beek NA, Wasserstein M, Zivkovic SA. A randomized study of alglucosidase alfa in late-onset Pompe's disease. N Engl J Med. 2010 Apr 15;362(15):1396-406. doi: 10.1056/NEJMoa0909859. PMID 20393176
- [Background] Slonim AE, Bulone L, Goldberg T, Minikes J, Slonim E, Galanko J, Martiniuk F. Modification of the natural history of adult-onset acid maltase deficiency by nutrition and exercise therapy. Muscle Nerve. 2007 Jan;35(1):70-7. doi: 10.1002/mus.20665. PMID 17022069
- [Background] Slonim AE, Coleman RA, McElligot MA, Najjar J, Hirschhorn K, Labadie GU, Mrak R, Evans OB, Shipp E, Presson R. Improvement of muscle function in acid maltase deficiency by high-protein therapy. Neurology. 1983 Jan;33(1):34-8. doi: 10.1212/wnl.33.1.34. PMID 6401355
- [Background] Kishnani PS, Steiner RD, Bali D, Berger K, Byrne BJ, Case LE, Crowley JF, Downs S, Howell RR, Kravitz RM, Mackey J, Marsden D, Martins AM, Millington DS, Nicolino M, O'Grady G, Patterson MC, Rapoport DM, Slonim A, Spencer CT, Tifft CJ, Watson MS. Pompe disease diagnosis and management guideline. Genet Med. 2006 May;8(5):267-88. doi: 10.1097/01.gim.0000218152.87434.f3. No abstract available. PMID 16702877
- [Background] Hagemans ML, Winkel LP, Van Doorn PA, Hop WJ, Loonen MC, Reuser AJ, Van der Ploeg AT. Clinical manifestation and natural course of late-onset Pompe's disease in 54 Dutch patients. Brain. 2005 Mar;128(Pt 3):671-7. doi: 10.1093/brain/awh384. Epub 2005 Jan 19. PMID 15659425
- [Background] Cupler EJ, Berger KI, Leshner RT, Wolfe GI, Han JJ, Barohn RJ, Kissel JT; AANEM Consensus Committee on Late-onset Pompe Disease. Consensus treatment recommendations for late-onset Pompe disease. Muscle Nerve. 2012 Mar;45(3):319-33. doi: 10.1002/mus.22329. Epub 2011 Dec 15. PMID 22173792
- [Background] Laforet P, Nicolino M, Eymard PB, Puech JP, Caillaud C, Poenaru L, Fardeau M. Juvenile and adult-onset acid maltase deficiency in France: genotype-phenotype correlation. Neurology. 2000 Oct 24;55(8):1122-8. doi: 10.1212/wnl.55.8.1122. PMID 11071489
- [Background] Wokke JH, Escolar DM, Pestronk A, Jaffe KM, Carter GT, van den Berg LH, Florence JM, Mayhew J, Skrinar A, Corzo D, Laforet P. Clinical features of late-onset Pompe disease: a prospective cohort study. Muscle Nerve. 2008 Oct;38(4):1236-45. doi: 10.1002/mus.21025. PMID 18816591
- [Background] Schoser B, Hill V, Raben N. Therapeutic approaches in glycogen storage disease type II/Pompe Disease. Neurotherapeutics. 2008 Oct;5(4):569-78. doi: 10.1016/j.nurt.2008.08.009. PMID 19019308
- [Background] Scriver CR. The metabolic & molecular bases of inherited disease. 8th ed. ed. New York: McGraw-Hill; 2001.
- [Background] Hesselink RP, Wagenmakers AJ, Drost MR, Van der Vusse GJ. Lysosomal dysfunction in muscle with special reference to glycogen storage disease type II. Biochim Biophys Acta. 2003 Mar 20;1637(2):164-70. doi: 10.1016/s0925-4439(02)00229-6. PMID 12633905
- [Background] Jones HN, Crisp KD, Asrani P, Sloane R, Kishnani PS. Quantitative assessment of lingual strength in late-onset Pompe disease. Muscle Nerve. 2015 May;51(5):731-5. doi: 10.1002/mus.24523. Epub 2015 Jan 16. PMID 25399907
- [Background] van den Berg LE, Zandbergen AA, van Capelle CI, de Vries JM, Hop WC, van den Hout JM, Reuser AJ, Zillikens MC, van der Ploeg AT. Low bone mass in Pompe disease: muscular strength as a predictor of bone mineral density. Bone. 2010 Sep;47(3):643-9. doi: 10.1016/j.bone.2010.06.021. Epub 2010 Jun 25. PMID 20601298